CLINICAL TRIAL: NCT00682929
Title: Cannabis for Spasticity in Multiple Sclerosis: A Placebo-Controlled Study
Brief Title: Cannabis for Spasticity in Multiple Sclerosis
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Unable to complete subject recruitment
Sponsor: University of California, Davis (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 251429; MS Society Award # RG 3781-A-1 (Other Grant/Funding Number: MS Society)
Record Dates: First submitted 2008-05-19; First posted 2008-05-23 (Estimated); Results first posted 2018-05-18 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-04

CONDITIONS: Multiple Sclerosis
Keywords: cannabis; marijuana; Multiple Sclerosis; spasticity
MeSH Terms: conditions — Multiple Sclerosis; Marijuana Abuse; Muscle Spasticity | interventions — nabiximols; Dronabinol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1) Inhaled Cannabis (Active Comparator): Inhaled cannabis is compared to oral placebo.
  Interventions: Drug: Inhaled Cannabis; Drug: Oral Placebo
- 2) Oral THC (Active Comparator): Inhaled placebo is compared to oral THC.
  Interventions: Drug: Oral THC; Drug: Inhaled placebo
- 3) Placebo (Placebo Comparator): Inhaled placebo is compared to oral placebo.
  Interventions: Drug: Oral Placebo; Drug: Inhaled placebo

INTERVENTIONS:
Drug: Inhaled Cannabis — Participants will be instructed to smoke one cannabis cigarette, daily for 7 weeks.
  Other Names: Cannabis
  Arms: 1) Inhaled Cannabis
Drug: Oral THC — Participants will be instructed to take two 5 mg dronabinol tablets two hours prior to the inhaled medication, daily for 7 weeks.
  Other Names: dronabinol
  Arms: 2) Oral THC
Drug: Oral Placebo — Participants will be instructed to take two placebo tablets two hours prior to the inhaled medication, daily for 7 weeks.
  Other Names: placebo
  Arms: 1) Inhaled Cannabis; 3) Placebo
Drug: Inhaled placebo — Participants will be instructed to smoke one placebo cigarette, daily for 7 weeks.
  Other Names: placebo
  Arms: 2) Oral THC; 3) Placebo

SUMMARY:
The purpose of this study is to learn if the use of inhaled cannabis (marijuana) and oral cannabinoid (dronabinol, Marinol or THC, which is an active ingredient of marijuana) is safe and effective in reducing the symptoms of spasticity and tremor in patients with secondary-progressive or primary progressive multiple sclerosis.

DETAILED DESCRIPTION:
The treatment of MS is far from satisfactory. For acute attacks, high dose corticosteroids seem to reduce the duration of attacks and to reduce the likelihood of future attacks. Immunomodulatory agents, available in this disease over the last decade, reduce the frequency of severe attacks by about one third. The remainder of the treatments are symptomatic, aimed at reducing the disability already present.

Recent research into the CB1 and CB2 cannabinoid receptor systems suggest that cannabis may have the potential for affecting both the pathogenic mechanisms and the symptoms of MS. In light of the autoimmune hypothesis of the etiology of MS, THC could directly alter immune function in a manner that might reduce (or increase) the primary pathology of the disease.

Comparisons: Three treatment arms will be compared:

1. inhaled cannabis and oral placebo
2. inhaled placebo and oral THC
3. inhaled placebo and oral placebo

The effects of these agents analyzed at 3 weeks and 7 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of clinically definite multiple sclerosis as defined by Poser criteria
* Moderate or severe spasticity
* Age 21 or older
* Must live close to the Sacramento, CA area

Exclusion Criteria:

* Preexisting pulmonary conditions, including poorly controlled asthma, chronic bronchitis, emphysema, bronchiectasis, and other significant pulmonary disorders
* Preexisting cardiac conditions, including ischemic heart disease, congestive heart failure, and other significant cardiac disorders
* Inability to abstain from tobacco or marijuana smoking, or use of alcohol or sedative or hypnotic medications during the duration of the study
* Pre-existing dementia, mania, depression or schizophrenia or other poorly controlled psychiatric illness
* Past history of abuse of recreational drugs, including marijuana and alcohol in the last 12 months
* History of or currently meets DSM-IV criteria for dependence on cannabis
* Use of cannabis, marijuana, or THC in the last four weeks
* Preexisting dementia, mania, depression, or schizophrenia or other poorly controlled psychiatric illness
* Exacerbation of MS within 30 days prior to screening visit
* Current use of cyclophosphamide, mitoxantrone, or cladribine
* Arthritis, bony and soft tissue disorders interfering with spasticity measures
* Inability to provide informed consent
* Recent cannabis use of more than twice per week one month prior to study entry
* For females of child bearing potential, inability to comply with adequate contraception

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2004-04-14 (Actual); Primary Completion 2011-08-17 (Actual); Study Completion 2011-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Apperson, MD, PhD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period began in April 2004 and continued through 2016. Subjects were recruited from the UC Davis Neurology Clinic and through self-referrals.
Groups:
- 1) Inhaled Cannabis: Inhaled cannabis is compared to oral placebo.
  Inhaled Cannabis: 20 people will be enrolled in this arm of the study and will receive study drug for 7 weeks. Subjects in this arm of the study will be instructed to take their oral medication (placebo for this group) two and a half hours prior to the inhaled medication. Subjects will take two pills and smoke one cannabis cigarette, daily.
- 2) Oral THC: Inhaled placebo is compared to oral THC.
  Oral THC: 20 people will be enrolled in this arm of the study and will receive study drug for 7 weeks. Subjects in this arm of the study will be instructed to take their oral medication (two 5mg dronabinol tablets) two and a half hours prior to the inhaled medication (placebo for this group). Subjects will take two pills and smoke one cigarette, daily.
- 3) Placebo: Inhaled placebo is compared to oral placebo.
  Placebo: 20 people will be enrolled in this arm of the study and will receive study drug for 7 weeks. Subjects in this arm of the study will be instructed to take their oral medication (placebo) two and a half hours prior to the inhaled medication (placebo). Subjects will take two pills and smoke one cigarette, daily.
Period: Overall Study
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Started | 13 | 14 | 14
Completed | 7 | 9 | 12
Not Completed | 6 | 5 | 2
Not completed — Adverse Event | 4 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 1
Not completed — dosing compliance < 80% | 0 | 2 | 0
Not completed — lag in DEA renewal | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo | Total
Number analyzed (Participants) | 13 | 14 | 14 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 13 | 12 | 38
  >=65 years | 0 | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 8 | 20
  Male | 8 | 7 | 6 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 13 | 14 | 14 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 1 | 5
  White | 11 | 12 | 13 | 36
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 14 | 14 | 41

OUTCOME MEASURES:

1. Primary Outcome: Change From Week 0 to Week 3 in the Rate of Torque Increase, Flexion
Description: A modified servo-controlled torque motor system (Lido WorkSet II) was designed for this study to analyze the resistance to passive movement of the knee. It determines the amount of torque required to move the knee joint (without voluntary resistance) at high velocities (up to 200 degrees per second) and at slow velocities (as low as 10 degrees per second). The slow displacement torque is a measure of the passive resistance to movement (from the connective tissue and the non-contracting muscle) and the rapid displacement torques are the sum of the passive and active (involuntary) resistance. The active (involuntary) resistance is the result of the stretch reflex and correlates well with the clinical assessment of spasticity. The change was calculated by taking the value at Week 3 and subtracting the value at Week 0. A negative result indicates a decrease in the torque measured and correlates to a decrease in spasticity and a better outcome.
Time Frame: Week 0, Week 3
Population: Only 28 subjects completed the study through the Wk 7 visit; 2 subjects who discontinued early (AE and withdraw by subject) were active at the Wk 3 visit and were included in the Wk 3 analysis; only 25 total subjects had Lido assessments at both the Week 0 and Week 3 study visits and were able to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: degrees/second
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 7 | 9 | 9
degrees/second | 0.0018 (0.0071) | -0.0121 (0.0183) | 0.0007 (0.0064)

2. Secondary Outcome: Change From Week 0 to Week 3 in Modified Ashworth Score (MAS)
Description: The Modified Ashworth scale measures resistance during passive soft-tissue stretching. Spasticity is graded on a scale of 0 (no increase in muscle tone) to 4 (affected part rigid in flexion or extension). The highest score (flexion or extension), for the lower extremities only, was used for each subject. The change was calculated by taking the Week 3 score and subtracting the Week 0 score. A negative result indicates a decrease in spasticity and correlates to a better outcome.
Time Frame: Week 0, Week 3
Population: Only 28 subjects completed the study through the Wk 7 visit; 2 subjects who discontinued early (AE and withdraw by subject) were active at the Wk 3 visit and were included in the Wk 3 analysis; 28 total subjects had Ashworth assessments at both the Week 0 and Week 3 study visits and were able to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 6 | 11 | 11
units on scale | -0.333 (1.0328) | 0 (0.8944) | -0.4545 (1.0357)

3. Secondary Outcome: Change From Week 0 to Week 7 in Modified Ashworth Score
Description: The Modified Ashworth scale measures resistance during passive soft-tissue stretching. Spasticity is graded on a scale of 0 (no increase in muscle tone) to 4 (affected part rigid in flexion or extension). The highest score (flexion or extension), for the lower extremities only, was used for each subject. The change was calculated by taking the Week 7 score and subtracting the Week 0 score. A negative result indicates a decrease in spasticity and correlates to a better outcome.
Time Frame: Week 0, Week 7
Population: Only 28 subjects completed the study through the Wk 7 visit; Of these 28 subjects, only 27 subjects had Ashworth assessments at both the Week 0 and Week 7 study visits and were able to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 7 | 8 | 12
units on a scale | 1.1429 (0.6901) | -0.3750 (0.5175) | -0.2500 (0.7538)

4. Secondary Outcome: Change From Week 0 to Week 3 in Ambulation Index (AI) Score
Description: The AI is a 9-point rating scale used to assess mobility by evaluating the time and degree of assistance required to walk 25 feet. Scores range from 0 (asymptomatic, fully active) to 9 (restricted to wheelchair, unable to transfer self independently). Lower scores represent a better outcome for MS patients. For this study, the AI score was based on the results of the 25 Foot Walk test, also performed at the study visit. The change was calculated by taking the Week 3 score and subtracting the Week 0 score. A negative result for this outcome indicates an improvement in ambulation and correlates to a better outcome.
Time Frame: Week 0, Week 3
Population: Only 28 subjects completed the study through the Wk 7 visit; 2 subjects who discontinued early (AE and withdraw by subject) were active at the Wk 3 visit and were included in the Wk 3 analysis; 27 total subjects had Ambulation Index assessments at both the Week 0 and Week 3 study visits and were able to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 6 | 10 | 11
units on a scale | 0 (0.6325) | 0 (0.6667) | 0.1818 (0.4045)

5. Secondary Outcome: Change From Week 0 to Week 7 in Ambulation Index (AI) Score
Description: The AI is a 9-point rating scale used to assess mobility by evaluating the time and degree of assistance required to walk 25 feet. Scores range from 0 (asymptomatic, fully active) to 9 (restricted to wheelchair, unable to transfer self independently). Lower scores represent a better outcome for MS patients. For this study, the AI score was based on the results of the 25 Foot Walk test, also performed at the study visit. The change was calculated by taking the Week 7 score and subtracting the Week 0 score. A negative result for this outcome indicates an improvement in ambulation and correlates to a better outcome.
Time Frame: Week 0, Week 7
Population: Only 28 subjects completed the study through the Wk 7 visit; Of these 28 subjects, all 28 subjects had Ambulation Index assessments at both the Week 0 and Week 7 study visits and were able to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 7 | 9 | 12
units on a scale | 0.1429 (0.3780) | 0.4444 (0.5270) | 0.3333 (0.6513)

6. Secondary Outcome: Change From Week 0 to Week 3 in 25 Foot Walk Time
Description: The Timed 25 Foot Walk is a quantitative measure of lower extremity function. The patient is instructed to walk on a marked 25-foot course, as quickly and as safely as possible. The patient is allowed to use his/her typical walking aid, if applicable. The task is completed twice and the average time of the two trials was used for this outcome measure. The change was calculated by taking the Week 3 time and subtracting the Week 0 time. A negative result indicates an improvement in walking ability and correlates to a better outcome.
Time Frame: Week 0, Week 3
Population: Only 28 subjects completed the study through the Wk 7 visit; 2 subjects who discontinued early (AE and withdraw by subject) were active at the Wk 3 visit and were included in the Wk 3 analysis; 22 total subjects had 25 Foot Walk tests performed at both the Week 0 and Week 3 study visits and were able to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 5 | 7 | 10
seconds | -0.0100 (1.6300) | -3.3714 (4.5605) | 0.1400 (1.9998)

7. Secondary Outcome: Change From Week 0 to Week 7 in 25 Foot Walk Time
Description: The Timed 25 Foot Walk is a quantitative measure of lower extremity function. The patient is instructed to walk on a marked 25-foot course, as quickly and as safely as possible. The patient is allowed to use his/her typical walking aid, if applicable. The task is completed twice and the average time of the two trials was used for this outcome measure. The change was calculated by taking the Week 7 time and subtracting the Week 0 time. A negative result indicates an improvement in walking ability and correlates to a better outcome.
Time Frame: Week 0, Week 7
Population: Only 28 subjects completed the study through the Wk 7 visit; Of these 28 subjects, only 26 subjects had 25 Foot Walk tests performed at both the Week 0 and Week 7 study visits and were able to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 6 | 9 | 11
seconds | -2.6000 (5.6240) | 3.3667 (9.7660) | 2.2773 (6.3507)

8. Primary Outcome: Change From Week 0 to Week 3 in the Rate of Torque Increase, Extension
Description: as for outcome 1
Time Frame: Week 0, Week 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: degrees/second
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 7 | 9 | 9
degrees/second | 0.0004 (0.0136) | -0.0310 (0.0780) | 0.0105 (0.0208)

9. Primary Outcome: Change From Week 0 to Week 7 in the Rate of Torque Increase, Flexion
Description: A modified servo-controlled torque motor system (Lido WorkSet II) was designed for this study to analyze the resistance to passive movement of the knee. It determines the amount of torque required to move the knee joint (without voluntary resistance) at high velocities (up to 200 degrees per second) and at slow velocities (as low as 10 degrees per second). The slow displacement torque is a measure of the passive resistance to movement (from the connective tissue and the non-contracting muscle) and the rapid displacement torques are the sum of the passive and active (involuntary) resistance. The active (involuntary) resistance is the result of the stretch reflex and correlates well with the clinical assessment of spasticity. The change was calculated by taking the value at Week 7 and subtracting the value at Week 0. A negative result indicates a decrease in the torque measured and correlates to a decrease in spasticity and a better outcome.
Time Frame: Week 0, Week 7
Population: Only 28 subjects completed the study through the Wk 7 visit; Of these 28 subjects, only 26 subjects had Lido assessments at both the Week 0 and Week 7 study visits and were able to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: degrees/second
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 7 | 8 | 11
degrees/second | -0.0013 (0.0405) | -0.0015 (0.0235) | 0.0043 (0.0161)

10. Primary Outcome: LIDO Machine Score - Rate of Torque Increase, Extension
Description: as for outcome 9
Time Frame: Week 0, Week 7
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: degrees/second
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 7 | 8 | 11
degrees/second | -0.0122 (0.0049) | -0.0019 (0.0256) | 0.0186 (0.0240)

11. Secondary Outcome: Change From Week 0 to Week 3 in 9 Hole Peg Test (Dominant Hand) Time
Description: The 9 hold peg test is a quantitative measure of upper extremity (arm and hand function). Patients are instructed to fill an 9 hole peg board with 1 peg at a time and then immediately remove the pegs, 1 at a time. The dominant hand is tested twice and the average time was used for this outcome measure. The change was calculated by taking the Week 3 time and subtracting the Week 0 time.
  A negative result indicates an improvement in arm and hand function and correlates with a better outcome.
Time Frame: Week 0, Week 3
Population: Only 28 subjects completed the study through the Wk 7 visit; 2 subjects who discontinued early (AE and withdraw by subject) were active at the Wk 3 visit and were included in the Wk 3 analysis; 26 total subjects had 9 Hole Peg tests (dominant hand) at both the Week 0 and Week 3 study visits and were able to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 7 | 9 | 10
seconds | -0.8929 (3.2680) | -1.5244 (7.8972) | 1.4450 (8.7548)

12. Secondary Outcome: Change From Week 0 to Week 7 in 9 Hole Peg Test (Dominant Hand) Time
Description: The 9 hold peg test is a quantitative measure of upper extremity (arm and hand function). Patients are instructed to fill an 9 hole peg board with 1 peg at a time and then immediately remove the pegs, 1 at a time. The dominant hand is tested twice and the average time was used for this outcome measure. The change was calculated by taking the Week 7 time and subtracting the Week 0 time.
  A negative result indicates an improvement in arm and hand function and correlates with a better outcome.
Time Frame: Week 0, Week 7
Population: Only 28 subjects completed the study through the Wk 7 visit; Of these 28 subjects, only 27 subjects had 9 Hole Peg tests (dominant hand) performed at both the Week 0 and Week 7 study visits and were able to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 7 | 9 | 11
seconds | 5.6714 (20.9260) | 1.4756 (11.3974) | -0.4991 (7.2244)

13. Secondary Outcome: Change From Week 0 to Week 3 in 9 Hole Peg Test (Non- Dominant Hand) Time
Description: The 9 hold peg test is a quantitative measure of upper extremity (arm and hand function). Patients are instructed to fill an 9 hole peg board with 1 peg at a time and then immediately remove the pegs, 1 at a time. The non-dominant hand is tested twice and the average time was used for this outcome measure. The change was calculated by taking the Week 3 time and subtracting the Week 0 time.
  A negative result indicates an improvement in arm and hand function and correlates with a better outcome.
Time Frame: Week 0, Week 3
Population: Only 28 subjects completed the study through the Wk 7 visit; 2 subjects who discontinued early (AE and withdraw by subject) were active at the Wk 3 visit and were included in the Wk 3 analysis; 26 total subjects had 9 Hole peg tests (non-dom. hand) at both the Week 0 and Week 3 study visits and were able to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 6 | 11 | 9
seconds | -1.0250 (2.5514) | 2.1318 (10.7380) | -1.3933 (3.0505)

14. Secondary Outcome: Change From Week 0 to Week 7 in 9 Hole Peg Test (Non- Dominant Hand) Time
Description: as for outcome 12
Time Frame: Week 0, Week 7
Population: Only 28 subjects completed the study through the Wk 7 visit; Of these 28 subjects, only 25 subjects had 9 Hole Peg tests (non-dom. hand) performed at both the Week 0 and Week 7 study visits and were able to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 6 | 9 | 10
seconds | -2.1083 (1.3786) | -3.9556 (10.5019) | 0.5530 (4.8470)

15. Secondary Outcome: Change From Week 0 to Week 3 in Paced Auditory Serial Addition Test (PASAT) Score
Description: The PASAT is a measure of cognitive function that specifically assesses auditory information processing speed and flexibility, as well as calculation ability; The test is presented via recording on a CD to control the rate of stimulus presentation. Single digits are presented every 3 seconds and the patient must add each new digit to the one immediately prior to it. The test score is the number of correct sums given (out of a possible 60) in each trial. There are 2 test forms, A and B. The forms were alternated and at least 1 practice test (10 sums) was performed prior to each trial. The change was calculated by taking the Week 3 score and subtracting the Week 0 score. A negative result indicates an improvement in performance and correlates with a better outcome.
Time Frame: Week 0, Week 3
Population: Only 28 subjects completed the study through the Wk 7 visit; 2 subjects who discontinued early (AE and withdraw by subject) were active at the Wk 3 visit and were included in the Wk 3 analysis; 29 total subjects had PASAT assessments at both the Week 0 and Week 3 study visits and were able to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: number correct
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 7 | 11 | 11
number correct | -3.7143 (10.0285) | 0.3636 (6.0212) | 2.5455 (8.8472)

16. Secondary Outcome: Change From Week 0 to Week 7 in Paced Auditory Serial Addition Test (PASAT) Score
Description: The PASAT is a measure of cognitive function that specifically assesses auditory information processing speed and flexibility, as well as calculation ability; The test is presented via recording on a CD to control the rate of stimulus presentation. Single digits are presented every 3 seconds and the patient must add each new digit to the one immediately prior to it. The test score is the number of correct sums given (out of a possible 60) in each trial. There are 2 test forms, A and B. The forms were alternated and at least 1 practice test (10 sums) was performed prior to each trial. The change was calculated by taking the Week 7 score and subtracting the Week 0 score. A negative result indicates an improvement in performance and correlates with a better outcome.
Time Frame: Week 0, Week 7
Population: Only 28 subjects completed the study through the Wk 7 visit; Of these 28 subjects, all 28 subjects had PASAT assessments at both the Week 0 and Week 7 study visits and were able to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: number correct
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 7 | 9 | 12
number correct | 2.0 (6.3770) | 0.1111 (5.6887) | 7.9167 (6.1120)

17. Secondary Outcome: Change From Week 0 to Week 3 in Functional System Score - Vision
Description: The EDSS is a method of quantifying disability in MS patients and monitoring changes in the level of disability over time. The EDSS quantifies disability in 7 functional systems (FS): visual, brainstem, pyramidal, cerebellar, sensory, bowel and bladder, and cerebral, and includes a measure of ambulation. Neurostatus version 10/2002 was used for this study. The FS Vision score is determined by a 7-point scale, with 0 being the lowest (normal) and 6 being the highest (grade 5 plus maximal visual acuity of better eye of 20/60 (0.3) or less).
  Higher values indicate more impaired vision. The change was calculated by taking the Week 3 score and subtracting the Week 0 score. A negative result indicates an improvement in vision and correlates to a better outcome.
Time Frame: Week 0, Week 3
Population: Only 28 subjects completed the study through the Wk 7 visit; 2 subjects who discontinued early (AE and withdraw by subject) were active at the Wk 3 visit and were included in the Wk 3 analysis; 27 total subjects had FS Vision assessments at both the Week 0 and Week 3 study visits and were able to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 6 | 10 | 11
units on a scale | 0.1667 (0.4082) | -0.3000 (0.2517) | -1.0 (0.6325)

18. Secondary Outcome: Change From Week 0 to Week 7 in Functional System Score - Vision
Description: The EDSS is a method of quantifying disability in MS patients and monitoring changes in the level of disability over time. The EDSS quantifies disability in 7 functional systems (FS): visual, brainstem, pyramidal, cerebellar, sensory, bowel and bladder, and cerebral, and includes a measure of ambulation. Neurostatus version 10/2002 was used for this study. The FS Vision score is determined by a 7-point scale, with 0 being the lowest (normal) and 6 being the highest (grade 5 plus maximal visual acuity of better eye of 20/60 (0.3) or less).
  Higher values indicate more impaired vision. The change was calculated by taking the Week 7 score and subtracting the Week 0 score. A negative result indicates an improvement in vision and correlates to a better outcome.
Time Frame: Week 0, Week 7
Population: Only 28 subjects completed the study through the Wk 7 visit; Of these 28 subjects, only 27 subjects had FS Vision assessments at both the Week 0 and Week 7 study visits and were able to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 7 | 8 | 12
units on a scale | -0.1429 (0.6901) | -0.3750 (0.9161) | -0.6667 (0.8876)

19. Secondary Outcome: Change From Week 0 to Week 3 in Functional System Score - Brainstem
Description: The EDSS is a method of quantifying disability in MS patients and monitoring changes in the level of disability over time. The EDSS quantifies disability in 7 functional systems (FS): visual, brainstem, pyramidal, cerebellar, sensory, bowel and bladder, and cerebral, and includes a measure of ambulation. Neurostatus version 10/2002 was used for this study. The FS Brainstem score is determined by a 6-point scale, with 0 being the lowest (normal) and 5 being the highest (inability to swallow or speak). Higher values indicate more impaired function. The change was calculated by taking the Week 3 score and subtracting the Week 0 score. A negative result indicates an improvement in function and correlates to a better outcome.
Time Frame: Week 0, Week 3
Population: Only 28 subjects completed the study through the Wk 7 visit; 2 subjects who discontinued early (AE and withdraw by subject) were active at the Wk 3 visit and were included in the Wk 3 analysis; 28 total subjects had FS Brainstem assessments at both the Week 0 and Week 3 study visits and were able to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 6 | 11 | 11
units on a scale | 0.1667 (0.4082) | -0.0909 (0.8312) | 0.2727 (1.4206)

20. Secondary Outcome: Change From Week 0 to Week 7 in Functional System Score - Brainstem
Description: The EDSS is a method of quantifying disability in MS patients and monitoring changes in the level of disability over time. The EDSS quantifies disability in 7 functional systems (FS): visual, brainstem, pyramidal, cerebellar, sensory, bowel and bladder, and cerebral, and includes a measure of ambulation. Neurostatus version 10/2002 was used for this study. The FS Brainstem score is determined by a 6-point scale, with 0 being the lowest (normal) and 5 being the highest (inability to swallow or speak). Higher values indicate more impaired function. The change was calculated by taking the Week 7 score and subtracting the Week 0 score. A negative result indicates an improvement in function and correlates to a better outcome.
Time Frame: Week 0, Week 7
Population: Only 28 subjects completed the study through the Wk 7 visit; Of these 28 subjects, only 27 subjects had FS Brainstem assessments at both the Week 0 and Week 7 study visits and were able to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 7 | 8 | 12
units on a scale | -0.1429 (0.6901) | 0.6250 (1.0607) | 0.1667 (1.0299)

21. Secondary Outcome: Change From Week 0 to Week 3 in Functional System Score - Pyramidal
Description: The EDSS is a method of quantifying disability in MS patients and monitoring changes in the level of disability over time. The EDSS quantifies disability in 7 functional systems (FS): visual, brainstem, pyramidal, cerebellar, sensory, bowel and bladder, and cerebral, and includes a measure of ambulation. Neurostatus version 10/2002 was used for this study. The FS Pyramidal score is determined by a 7-point scale, with 0 being the lowest (normal) and 6 being the highest (tetraplegia (grade 0 or 1 in all muscle groups of upper and lower limbs). Higher values indicate more impaired function. The change was calculated by taking the Week 3 score and subtracting the Week 0 score. A negative result indicates an improvement in function and correlates to a better outcome.
Time Frame: Week 0, Week 3
Population: Only 28 subjects completed the study through the Wk 7 visit; 2 subjects who discontinued early (AE and withdraw by subject) were active at the Wk 3 visit and were included in the Wk 3 analysis; 28 total subjects had FS Pyramidal assessments at both the Week 0 and Week 3 study visits and were able to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 6 | 11 | 11
units on a scale | 0.3333 (1.2111) | -0.1818 (0.6030) | 0 (0.6325)

22. Secondary Outcome: Change From Week 0 to Week 7 in Functional System Score - Pyramidal
Description: The EDSS is a method of quantifying disability in MS patients and monitoring changes in the level of disability over time. The EDSS quantifies disability in 7 functional systems (FS): visual, brainstem, pyramidal, cerebellar, sensory, bowel and bladder, and cerebral, and includes a measure of ambulation. Neurostatus version 10/2002 was used for this study. The FS Pyramidal score is determined by a 7-point scale, with 0 being the lowest (normal) and 6 being the highest (tetraplegia (grade 0 or 1 in all muscle groups of upper and lower limbs). Higher values indicate more impaired function. The change was calculated by taking the Week 7 score and subtracting the Week 0 score. A negative result indicates an improvement in function and correlates to a better outcome.
Time Frame: Week 0, Week 7
Population: Only 28 subjects completed the study through the Wk 7 visit; Of these 28 subjects, only 27 subjects had FS Pyramidal assessments at both the Week 0 and Week 7 study visits and were able to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 7 | 8 | 12
units on a scale | 0.4286 (0.9759) | -0.5000 (1.0690) | 0.0833 (0.6686)

23. Secondary Outcome: Change From Week 0 to Week 3 in Functional System Score - Cerebellar
Description: The EDSS is a method of quantifying disability in MS patients and monitoring changes in the level of disability over time. The EDSS quantifies disability in 7 functional systems (FS): visual, brainstem, pyramidal, cerebellar, sensory, bowel and bladder, and cerebral, and includes a measure of ambulation. Neurostatus version 10/2002 was used for this study. The FS Cerebellar score is determined by a 6-point scale, with 0 being the lowest (normal) and 5 being the highest (unable to perform coordinated movements due to ataxia). Higher values indicate more impaired function. The change was calculated by taking the Week 3 score and subtracting the Week 0 score. A negative result indicates an improvement in function and correlates to a better outcome.
Time Frame: Week 0, Week 3
Population: Only 28 subjects completed the study through the Wk 7 visit; 2 subjects who discontinued early (AE and withdraw by subject) were active at the Wk 3 visit and were included in the Wk 3 analysis; 27 total subjects had FS Cerebellar assessments at both the Week 0 and Week 3 study visits and were able to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 6 | 10 | 11
units on a scale | -0.50 (0.5477) | -0.20 (0.9189) | -0.0909 (0.5394)

24. Secondary Outcome: Change From Week 0 to Week 7 in Functional System Score - Cerebellar
Description: The EDSS is a method of quantifying disability in MS patients and monitoring changes in the level of disability over time. The EDSS quantifies disability in 7 functional systems (FS): visual, brainstem, pyramidal, cerebellar, sensory, bowel and bladder, and cerebral, and includes a measure of ambulation. Neurostatus version 10/2002 was used for this study. The FS Cerebellar score is determined by a 6-point scale, with 0 being the lowest (normal) and 5 being the highest (unable to perform coordinated movements due to ataxia). Higher values indicate more impaired function. The change was calculated by taking the Week 7 score and subtracting the Week 0 score. A negative result indicates an improvement in function and correlates to a better outcome.
Time Frame: Week 0, Week 7
Population: Only 28 subjects completed the study through the Wk 7 visit; Of these 28 subjects, only 27 subjects had FS Cerebellar assessments at both the Week 0 and Week 7 study visits and were able to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 7 | 8 | 12
units on a scale | -0.5714 (0.7868) | -0.7500 (0.7071) | 0.0 (1.2792)

25. Secondary Outcome: Change From Week 0 to Week 3 in Functional System Score - Sensory
Description: The EDSS is a method of quantifying disability in MS patients and monitoring changes in the level of disability over time. The EDSS quantifies disability in 7 functional systems (FS): visual, brainstem, pyramidal, cerebellar, sensory, bowel and bladder, and cerebral, and includes a measure of ambulation. Neurostatus version 10/2002 was used for this study. The FS Sensory score is determined by a 7-point scale, with 0 being the lowest (normal) and 6 being the highest (sensation essentially lost below the head). Higher values indicate more impaired function. The change was calculated by taking the Week 3 score and subtracting the Week 0 score. A negative result indicates an improvement in function and correlates to a better outcome.
Time Frame: Week 0, Week 3
Population: Only 28 subjects completed the study through the Wk 7 visit; 2 subjects who discontinued early (AE and withdraw by subject) were active at the Wk 3 visit and were included in the Wk 3 analysis; 28 total subjects had FS Sensory assessments at both the Week 0 and Week 3 study visits and were able to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 6 | 11 | 11
units on a scale | -0.1667 (0.7528) | 0.0 (0.7746) | -0.1818 (1.3280)

26. Secondary Outcome: Change From Week 0 to Week 7 in Functional System Score - Sensory
Description: The EDSS is a method of quantifying disability in MS patients and monitoring changes in the level of disability over time. The EDSS quantifies disability in 7 functional systems (FS): visual, brainstem, pyramidal, cerebellar, sensory, bowel and bladder, and cerebral, and includes a measure of ambulation. Neurostatus version 10/2002 was used for this study. The FS Sensory score is determined by a 7-point scale, with 0 being the lowest (normal) and 6 being the highest (sensation essentially lost below the head). Higher values indicate more impaired function. The change was calculated by taking the Week 7 score and subtracting the Week 0 score. A negative result indicates an improvement in function and correlates to a better outcome.
Time Frame: Week 0, Week 7
Population: Only 28 subjects completed the study through the Wk 7 visit; Of these 28 subjects, only 27 subjects had FS Sensory assessments at both the Week 0 and Week 7 study visits and were able to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 7 | 8 | 12
units on a scale | 0.0 (0.8165) | -0.1250 (1.4577) | -0.3333 (1.8749)

27. Secondary Outcome: Change From Week 0 to Week 3 in Functional System Score - Bowel and Bladder
Description: The EDSS is a method of quantifying disability in MS patients and monitoring changes in the level of disability over time. The EDSS quantifies disability in 7 functional systems (FS): visual, brainstem, pyramidal, cerebellar, sensory, bowel and bladder, and cerebral, and includes a measure of ambulation. Neurostatus version 10/2002 was used for this study. The FS Bowel and Bladder score is determined by a 7-point scale, with 0 being the lowest (normal) and 6 being the highest (loss of bowel and bladder function). Higher values indicate more impaired function. The change was calculated by taking the Week 3 score and subtracting the Week 0 score. A negative result indicates an improvement in function and correlates to a better outcome.
Time Frame: Week 0, Week 3
Population: Only 28 subjects completed the study through the Wk 7 visit; 2 subjects who discontinued early (AE and withdraw by subject) were active at the Wk 3 visit and were included in the Wk 3 analysis; 28 total subjects had FS Bowel & Bladder assessments at both the Week 0 and Week 3 study visits and were able to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 6 | 11 | 11
units on a scale | -0.1667 (0.4082) | 0.0 (1.0954) | -0.2727 (1.1909)

28. Secondary Outcome: Change From Week 0 to Week 7 in Functional System Score - Bowel and Bladder
Description: The EDSS is a method of quantifying disability in MS patients and monitoring changes in the level of disability over time. The EDSS quantifies disability in 7 functional systems (FS): visual, brainstem, pyramidal, cerebellar, sensory, bowel and bladder, and cerebral, and includes a measure of ambulation. Neurostatus version 10/2002 was used for this study. The FS Bowel and Bladder score is determined by a 7-point scale, with 0 being the lowest (normal) and 6 being the highest (loss of bowel and bladder function). Higher values indicate more impaired function. The change was calculated by taking the Week 7 score and subtracting the Week 0 score. A negative result indicates an improvement in function and correlates to a better outcome.
Time Frame: Week 0, Week 7
Population: Only 28 subjects completed the study through the Wk 7 visit; Of these 28 subjects, only 27 subjects had FS Bowel & Bladder assessments at both the Week 0 and Week 7 study visits and were able to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 7 | 8 | 12
units on a scale | -0.5714 (1.1339) | 0.2500 (1.2817) | -0.3333 (1.1547)

29. Secondary Outcome: Change From Week 0 to Week 3 in Functional System Score - Cerebral
Description: The EDSS is a method of quantifying disability in MS patients and monitoring changes in the level of disability over time. The EDSS quantifies disability in 7 functional systems (FS): visual, brainstem, pyramidal, cerebellar, sensory, bowel and bladder, and cerebral, and includes a measure of ambulation. Neurostatus version 10/2002 was used for this study. The FS Cerebral score is determined by a 6-point scale, with 0 being the lowest (normal) and 5 being the highest (dementia). Higher values indicate more impaired function. The change was calculated by taking the Week 3 score and subtracting the Week 0 score. A negative result indicates an improvement in function and correlates to a better outcome. Fatigue did not contribute to this FS score or the EDSS total score.
Time Frame: Week 0, Week 3
Population: Only 28 subjects completed the study through the Wk 7 visit; 2 subjects who discontinued early (AE and withdraw by subject) were active at the Wk 3 visit and were included in the Wk 3 analysis; 28 total subjects had FS Cerebral assessments at both the Week 0 and Week 3 study visits and were able to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 6 | 11 | 11
units on a scale | 0.50 (0.8367) | 0.0 (0.6325) | -0.3636 (0.8090)

30. Secondary Outcome: Change From Week 0 to Week 7 in Functional System Score - Cerebral
Description: The EDSS is a method of quantifying disability in MS patients and monitoring changes in the level of disability over time. The EDSS quantifies disability in 7 functional systems (FS): visual, brainstem, pyramidal, cerebellar, sensory, bowel and bladder, and cerebral, and includes a measure of ambulation. Neurostatus version 10/2002 was used for this study. The FS Cerebral score is determined by a 6-point scale, with 0 being the lowest (normal) and 5 being the highest (dementia). Higher values indicate more impaired function. The change was calculated by taking the Week 7 score and subtracting the Week 0 score. A negative result indicates an improvement in function and correlates to a better outcome. Fatigue did not contribute to this FS score or the EDSS total score.
Time Frame: Week 0, Week 7
Population: Only 28 subjects completed the study through the Wk 7 visit; Of these 28 subjects, only 27 subjects had FS Cerebral assessments at both the Week 0 and Week 7 study visits and were able to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 7 | 8 | 12
units on a scale | 0.4286 (0.5345) | 0.0 (0.5345) | -0.2500 (0.8660)

31. Secondary Outcome: Change From Week 0 to Week 3 in Expanded Disability Status Score (EDSS)
Description: The EDSS is a method of quantifying disability in MS patients and monitoring changes in the level of disability over time. The EDSS quantifies disability in 7 functional systems (FS): visual, brainstem, pyramidal, cerebellar, sensory, bowel and bladder, and cerebral, and includes a measure of ambulation. Neurostatus version 10/2002 was used for this study. The total EDSS score ranges from 0 to 10, in 0.5 unit increments. A score of 0 is the lowest (normal neurological exam) and 10 is the highest (death due to MS). Higher values indicate more impaired function. The change was calculated by taking the Week 3 score and subtracting the Week 0 score. A negative result indicates an improvement in function and correlates to a better outcome.
Time Frame: Week 0, Week 3
Population: Only 28 subjects completed the study through the Wk 7 visit; 2 subjects who discontinued early (AE and withdraw by subject) were active at the Wk 3 visit and were included in the Wk 3 analysis; 28 total subjects had completed & scored EDSS assessments at both the Week 0 and Week 3 study visits and were able to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 6 | 11 | 11
units on a scale | -0.0833 (0.2041) | 0.0909 (0.3015) | -0.2727 (0.5641)

32. Secondary Outcome: Change From Week 0 to Week 7 in Expanded Disability Status Score (EDSS)
Description: The EDSS is a method of quantifying disability in MS patients and monitoring changes in the level of disability over time. The EDSS quantifies disability in 7 functional systems (FS): visual, brainstem, pyramidal, cerebellar, sensory, bowel and bladder, and cerebral, and includes a measure of ambulation. Neurostatus version 10/2002 was used for this study. The total EDSS score ranges from 0 to 10, in 0.5 unit increments. A score of 0 is the lowest (normal neurological exam) and 10 is the highest (death due to MS). Higher values indicate more impaired function. The change was calculated by taking the Week 7 score and subtracting the Week 0 score. A negative result indicates an improvement in function and correlates to a better outcome.
Time Frame: Week 0, Week 7
Population: Only 28 subjects completed the study through the Wk 7 visit; Of these 28 subjects, only 27 subjects had completed & scored EDSS assessments at both the Week 0 and Week 7 study visits and were able to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 7 | 8 | 12
units on a scale | 0.0714 (0.3450) | 0.0 (0.0) | -0.2083 (0.6557)

33. Secondary Outcome: Change From Week 0 to Week 3 in MS Quality of Life Inventory (MSQLI) - SF-36 Physical Component Score
Description: The SF-36 is a 36-item scale developed as a generic health status measure. It is a part of the MS Quality of Life Inventory. It can be reported as 2 summary scales - the Physical and Mental components. The scale is measured from 0 -100. The scale is set up so that a higher score indicates better health. The change was calculated by taking the Week 3 score and subtracting the Week 0 score. A positive result indicates an improvement in health status and correlates to a better outcome. A negative result indicates a decline in health and correlates to a worse outcome.
Time Frame: Week 0, Week 3
Population: Only 28 subjects completed the study through the Wk 7 visit; 2 subjects who discontinued early (AE & withdraw by subject) were active at the Wk 3 visit and were included in the Wk 3 analysis; 21 total subjects completed all SF-36 physical component questions at both the Wk 0 and Wk 3 study visits and were analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 7 | 7 | 7
units on a scale | 2.5734 (9.1669) | 4.3401 (9.9668) | 1.2656 (6.3093)

34. Secondary Outcome: Change From Week 0 to Week 7 in MS Quality of Life Inventory (MSQLI) - SF-36 Physical Component Score
Description: The SF-36 is a 36-item scale developed as a generic health status measure. It is a part of the MS Quality of Life Inventory. It can be reported as 2 summary scales - the Physical and Mental components. The scale is measured from 0 -100. The scale is set up so that a higher score indicates better health. The change was calculated by taking the Week 7 score and subtracting the Week 0 score. A positive result indicates an improvement in health status and correlates to a better outcome. A negative result indicates a decline in health and correlates to a worse outcome.
Time Frame: Week 0, Week 7
Population: Only 28 subjects completed the study through the Wk 7 visit; Of these 28 subjects, only 23 subjects completed all SF-36 physical component questions at both the Week 0 and Week 7 study visits and were able to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 6 | 7 | 10
units on a scale | -0.8695 (5.7636) | 1.0957 (7.9274) | -0.8803 (7.4724)

35. Secondary Outcome: Change From Week 0 to Week 3 in MS Quality of Life Inventory (MSQLI) - SF-36 Mental Component Score
Description: The SF-36 is a 36-item scale developed as a generic health status measure. It is a part of the MS Quality of Life Inventory. It can be reported as 2 summary scales - the Physical and Mental components. The scale is measured from 0 -100. The scale is set up so that a higher score indicates better health. The change was calculated by taking the Week 3 score and subtracting the Week 0. A positive result indicates an improvement in mental health status and correlates to a better outcome. A negative result indicates a decline in mental health and correlates to a worse outcome.
Time Frame: Week 0, Week 3
Population: Only 28 subjects completed the study through the Wk 7 visit; 2 subjects who discontinued early (AE & withdraw by subject) were active at the Wk 3 visit and were included in the Wk 3 analysis; 21 total subjects completed all SF-36 mental component questions at both the Wk 0 and Wk 3 study visits and were analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 7 | 7 | 7
units on a scale | 0.7606 (13.7458) | -4.3820 (9.6916) | 2.9471 (6.8578)

36. Secondary Outcome: Change From Week 0 to Week 7 in MS Quality of Life Inventory (MSQLI) - SF-36 Mental Component
Description: as for outcome 35
Time Frame: Week 0, Week 7
Population: Only 28 subjects completed the study through the Wk 7 visit; Of these 28 subjects, only 23 subjects completed all SF-36 mental component questions at both the Week 0 and Week 7 study visits and were able to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 6 | 7 | 10
units on a scale | 5.7328 (12.6299) | -2.0820 (13.4123) | 1.6035 (13.9515)

37. Secondary Outcome: Change From Week 0 to Week3 in MS Quality of Life Inventory (MSQLI) - Modified Fatigue Index Score
Description: The Modified Fatigue Index is a 21-item scale developed to assess the perceived impact of fatigue on daily activities. It is a part of the MS Quality of Life Inventory. The scale is measured from 0-84. The scale is set up so that a higher score indicates a greater impact of fatigue on a patient's daily activities. The change was calculated by taking the Week 3 score and subtracting the Week 0 score. A negative result indicates a decrease in the impact of fatigue on daily activities and correlates to a better outcome. A positive result indicates an increase in the impact of fatigue on daily activities and correlates to a worse outcome.
Time Frame: Week 0, Week 3
Population: Only 28 subjects completed the study through the Wk 7 visit; 2 subjects who discontinued early (AE & withdraw by subject) were active at the Wk 3 visit and were included in the Wk 3 analysis; 26 total subjects completed all Modified Fatigue Index questions at both the Wk 0 and Wk 3 study visits and were analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 6 | 10 | 10
units on a scale | -11.3333 (10.7641) | 1.2000 (10.9016) | -9.600 (16.5341)

38. Secondary Outcome: Change From Week 0 to Week 7 in MS Quality of Life Inventory (MSQLI) - Modified Fatigue Index Score
Description: The Modified Fatigue Index is a 21-item scale developed to assess the perceived impact of fatigue on daily activities. It is a part of the MS Quality of Life Inventory. The scale is measured from 0 - 84. The scale is set up so that a higher score indicates a greater impact of fatigue on a patient's daily activities. The change was calculated by taking the Week 7 score and subtracting the Week 0 score. A negative result indicates a decrease in the impact of fatigue on daily activities and correlates to a better outcome. A positive result indicates an increase in the impact of fatigue on daily activities and correlates to a worse outcome.
Time Frame: Week 0, Week 7
Population: Only 28 subjects completed the study through the Wk 7 visit; Of these 28 subjects, only 26 subjects completed all Modified Fatigue Index questions at both the Week 0 and Week 7 study visits and were able to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 6 | 9 | 11
units on a scale | -15.50 (11.3798) | 1.3333 (6.3836) | -11.0909 (18.4470)

39. Secondary Outcome: Change From Week 0 to Week 3 in MS Quality of Life Inventory (MSQLI) - Pain Effects Scale Score
Description: The Pain Effects Scale is a 6-item scale developed to assess the effects of pain on behavior and mood. It is a part of the MS Quality of Life Inventory. The scale is measured from 6-30. The scale is set up so that a higher score indicates a greater impact of pain on a patient's mood and behavior. The change was calculated by taking the Week 3 score and subtracting the Week 0 score. A negative result indicates a decrease in the impact of pain on mood and behavior and correlates to a better outcome. A positive result indicates an increase in the impact of pain on mood and behavior and correlates to a worse outcome.
Time Frame: Week 0, Week 3
Population: Only 28 subjects completed the study through the Wk 7 visit; 2 subjects who discontinued early (AE & withdraw by subject) were active at the Wk 3 visit and were included in the Wk 3 analysis; 28 total subjects completed all Pain Effects scale questions at both the Wk 0 and Wk 3 study visits and were analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 7 | 10 | 11
units on a scale | -1.0 (4.2032) | -2.20 (5.0067) | -2.5455 (5.8028)

40. Secondary Outcome: Change From Week 0 to Week 7 in MS Quality of Life Inventory (MSQLI) - Pain Effects Scale Score
Description: The Pain Effects Scale is a 6-item scale developed to assess the effects of pain on behavior and mood. It is a part of the MS Quality of Life Inventory. The scale is measured from 6-30. The scale is set up so that a higher score indicates a greater impact of pain on a patient's mood and behavior. The change was calculated by taking the Week 7 score and subtracting the Week 0 score. A negative result indicates a decrease in the impact of pain on mood and behavior and correlates to a better outcome. A positive result indicates an increase in the impact of pain on mood and behavior and correlates to a worse outcome.
Time Frame: Week 0, Week 7
Population: Only 28 subjects completed the study through the Wk 7 visit; Of these 28 subjects, all 28 subjects completed all Pain Effects scale questions at both the Week 0 and Week 7 study visits and were able to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 7 | 9 | 12
units on a scale | -2.5714 (5.9121) | -2.4444 (5.2228) | -2.500 (4.5627)

41. Secondary Outcome: Change From Week 0 to Week 3 in MS Quality of Life Inventory (MSQLI) - Sexual Satisfaction Scale Score
Description: The Sexual Satisfaction Scale is a 4-item scale developed to assess the impact of multiple sclerosis on sexual function and satisfaction. It is a part of the MS Quality of Life Inventory. The scale is measured from 4-24. The scale is set up so that a higher score indicates greater problems with sexual satisfaction. Subjects that answered "No" to the question, "Do you have a relationship with one primary partner", did not complete the scale. The change was calculated by taking the Week 3 score and subtracting the Week 0 score. A negative result indicates an improvement in sexual satisfaction and correlates to a better outcome. A positive result indicates a decrease in sexual satisfaction and correlates to a worse outcome.
Time Frame: Week 0, Week 3
Population: Only 28 subjects completed the study through the Wk 7 visit; 2 subjects who discontinued early (AE & withdraw by subject) were active at the Wk 3 visit and were included in the Wk 3 analysis; 19 total subjects completed all Sexual Satisfaction scale questions at both the Wk 0 and Wk 3 study visits and were analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 4 | 6 | 9
units on a scale | -4.250 (3.5940) | 0.6667 (0.8165) | -0.7778 (2.5386)

42. Secondary Outcome: Change From Week 0 to Week 7 in MS Quality of Life Inventory (MSQLI) - Sexual Satisfaction Scale Score
Description: The Sexual Satisfaction Scale is a 4-item scale developed to assess the impact of multiple sclerosis on sexual function and satisfaction. It is a part of the MS Quality of Life Inventory. The scale is measured from 4-24. The scale is set up so that a higher score indicates greater problems with sexual satisfaction. Subjects that answered "No" to the question, "Do you have a relationship with one primary partner", did not complete the scale. The change was calculated by taking the Week 7 score and subtracting the Week 0 score. A negative result indicates an improvement in sexual satisfaction and correlates to a better outcome. A positive result indicates a decrease in sexual satisfaction and correlates to a worse outcome.
Time Frame: Week 0, Week 7
Population: Only 28 subjects completed the study through the Wk 7 visit; Of these 28 subjects, only 19 subjects completed all Sexual Satisfaction scale questions at both the Week 0 and Week 7 study visits and were able to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 4 | 6 | 9
units on a scale | -3.750 (2.0616) | 0.1667 (3.1252) | 2.5556 (6.0438)

43. Secondary Outcome: Change From Week 0 to Week 3 in MS Quality of Life Inventory (MSQLI) - Bladder Control Scale Score
Description: The Bladder Control Scale is a 4-item scale developed to assess the impact of multiple sclerosis on bladder function. It is a part of the MS Quality of Life Inventory. The scale is measured from 0-22. The scale is set up so that a higher score indicates greater bladder control problems. The change was calculated by taking the Week 3 score and subtracting the Week 0 score. A negative result indicates an improvement in bladder control and correlates to a better outcome. A positive result indicates a decrease in bladder control and correlates to a worse outcome.
Time Frame: Week 0, Week 3
Population: Only 28 subjects completed the study through the Wk 7 visit; 2 subjects who discontinued early (AE & withdraw by subject) were active at the Wk 3 visit and were included in the Wk 3 analysis; 27 total subjects completed all Bladder Control scale questions at both the Wk 0 and Wk 3 study visits and were analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 6 | 10 | 11
units on a scale | 0.500 (2.0736) | -0.700 (6.3254) | -2.1818 (7.7951)

44. Secondary Outcome: Change From Week 0 to Week 7 in MS Quality of Life Inventory (MSQLI) - Bladder Control Scale Score
Description: The Bladder Control Scale is a 4-item scale developed to assess the impact of multiple sclerosis on bladder function. It is a part of the MS Quality of Life Inventory. The scale is measured from 0-22. The scale is set up so that a higher score indicates greater bladder control problems. The change was calculated by taking the Week 7 score and subtracting the Week 0 score. A negative result indicates an improvement in bladder control and correlates to a better outcome. A positive result indicates a decrease in bladder control and correlates to a worse outcome.
Time Frame: Week 0, Week 7
Population: Only 28 subjects completed the study through the Wk 7 visit; Of these 28 subjects, all 28 subjects completed all Bladder Control scale questions at both the Week 0 and Week 7 study visits and were able to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 7 | 9 | 12
units on a scale | -0.8571 (4.0999) | -1.8889 (5.2068) | -2.500 (6.0977)

45. Secondary Outcome: Change From Week 0 to Week 3 in MS Quality of Life Inventory (MSQLI) - Bowel Control Scale Score
Description: The Bowel Control Scale is a 5-item scale developed to assess the impact of multiple sclerosis on bowel function. It is a part of the MS Quality of Life Inventory. The scale is measured from 0-26. The scale is set up so that a higher score indicates greater bowel control problems. The change was calculated by taking the Week 3 score and subtracting the Week 0 score. A negative result indicates an improvement in bowel control and correlates to a better outcome. A positive result indicates a decrease in bowel control and correlates to a worse outcome.
Time Frame: Week 0, Week 3
Population: Only 28 subjects completed the study through the Wk 7 visit; 2 subjects who discontinued early (AE & withdraw by subject) were active at the Wk 3 visit and were included in the Wk 3 analysis; 26 total subjects completed all Bowel Control scale questions at both the Wk 0 and Wk 3 study visits and were analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 7 | 10 | 9
units on a scale | -0.7143 (4.4240) | -1.000 (4.8762) | 0.7778 (2.1667)

46. Secondary Outcome: Change From Week 0 to Week 7 in MS Quality of Life Inventory (MSQLI) - Bowel Control Scale Score
Description: The Bowel Control Scale is a 5-item scale developed to assess the impact of multiple sclerosis on bowel function. It is a part of the MS Quality of Life Inventory. The scale is measured from 0-26. The scale is set up so that a higher score indicates greater bowel control problems. The change was calculated by taking the Week 7 score and subtracting the Week 0 score. A negative result indicates an improvement in bowel control and correlates to a better outcome. A positive result indicates a decrease in bowel control and correlates to a worse outcome.
Time Frame: Week 0, Week 7
Population: Only 28 subjects completed the study through the Wk 7 visit; Of these 28 subjects, only 27 subjects completed all Bowel Control scale questions at both the Week 0 and Week 7 study visits and were able to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 7 | 9 | 11
units on a scale | -0.7143 (4.4615) | 0.2222 (2.7739) | 0.4545 (3.5599)

47. Secondary Outcome: Change From Week 0 to Week 3 in MS Quality of Life Inventory (MSQLI) - Impact of Visual Impairment Scale Score
Description: The Impact of Visual Impairment Scale is a 5-item scale developed to assess the extent to which activities dependent on vision are affected by MS-related visual problems. It is a part of the MS Quality of Life Inventory. The scale is measured from 0-15. The scale is set up so that a higher score indicates greater impact of visual problems on daily activities. The change was calculated by taking the Week 3 score and subtracting the Week 0 score. A negative result indicates a decrease in the impact of visual problems on daily activities and correlates to a better outcome. A positive result indicates an increase in the impact of visual problems on daily activities and correlates to a worse outcome.
Time Frame: Week 0, Week 3
Population: Only 28 subjects completed the study through the Wk 7 visit; 2 subjects who discontinued early (AE & withdraw by subject) were active at the Wk 3 visit and were included in the Wk 3 analysis; 27 total subjects completed all Impact of Visual Impairment scale questions at both the Wk 0 and Wk 3 study visits and were analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 7 | 9 | 11
units on a scale | -0.2857 (1.2536) | 0.5556 (1.6667) | 0.00 (2.5690)

48. Secondary Outcome: Change From Week 0 to Week 7 in MS Quality of Life Inventory (MSQLI) - Impact of Visual Impairment Scale Score
Description: The Impact of Visual Impairment Scale is a 5-item scale developed to assess the extent to which activities dependent on vision are affected by MS-related visual problems. It is a part of the MS Quality of Life Inventory. The scale is measured from 0-15. The scale is set up so that a higher score indicates greater impact of visual problems on daily activities. The change was calculated by taking the Week 7 score and subtracting the Week 0 score. A negative result indicates a decrease in the impact of visual problems on daily activities and correlates to a better outcome. A positive result indicates an increase in the impact of visual problems on daily activities and correlates to a worse outcome.
Time Frame: Week 0, Week 7
Population: Only 28 subjects completed the study through the Wk 7 visit; Of these 28 subjects, only 27 subjects completed all Impact of Visual Impairment scale questions at both the Week 0 and Week 7 study visits and were able to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 7 | 8 | 12
units on a scale | 0.5714 (0.7868) | 0.2500 (1.9821) | -0.7500 (1.7645)

49. Secondary Outcome: Change From Week 0 to Week 3 in MS Quality of Life Inventory (MSQLI) - Perceived Deficits Scale Score
Description: The Perceived Deficits Scale is a 20-item scale developed to assess the patient's perceived cognitive deficits. It is composed of four 5-item subscales: Attention/Concentration, Retrospective Memory, Prospective Memory, and Planning/Organization. It is a part of the MS Quality of Life Inventory. The total score is measured from 0-80. The scale is set up so that a higher score indicates greater perceived cognitive impairment. The change was calculated by taking the Week 3 score and subtracting the Week 0 score. A negative result indicates a decrease in the perception of cognitive impairment. A positive result indicates an increase in the perception of cognitive impairment. Since patient perceptions of cognitive impairment may not correlate with objective measures of cognitive impairment, the results should be interpreted with caution.
Time Frame: Week 0, Week 3
Population: Only 28 subjects completed the study through the Wk 7 visit; 2 subjects who discontinued early (AE & withdraw by subject) were active at the Wk 3 visit and were included in the Wk 3 analysis; 27 total subjects completed all Perceived Deficits scale questions at both the Wk 0 and Wk 3 study visits and were analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 7 | 10 | 10
units on a scale | -3.2857 (10.7659) | 3.000 (6.5828) | -6.600 (14.4929)

50. Secondary Outcome: Change From Week 0 to Week 7 in MS Quality of Life Inventory (MSQLI) - Perceived Deficits Scale Score
Description: The Perceived Deficits Scale is a 20-item scale developed to assess the patient's perceived cognitive deficits. It is composed of four 5-item subscales: Attention/Concentration, Retrospective Memory, Prospective Memory, and Planning/Organization. It is a part of the MS Quality of Life Inventory. The total score is measured from 0-80. The scale is set up so that a higher score indicates greater perceived cognitive impairment. The change was calculated by taking the Week 7 score and subtracting the Week 0 score. A negative result indicates a decrease in the perception of cognitive impairment. A positive result indicates an increase in the perception of cognitive impairment. Since patient perceptions of cognitive impairment may not correlate with objective measures of cognitive impairment, the results should be interpreted with caution.
Time Frame: Week 0, Week 7
Population: Only 28 subjects completed the study through the Wk 7 visit; Of these 28 subjects, only 26 subjects completed all Perceived Deficits scale questions at both the Week 0 and Week 7 study visits and were able to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 7 | 8 | 11
units on a scale | -4.8571 (13.0822) | 4.3750 (5.4494) | -2.0909 (10.2903)

51. Secondary Outcome: Change From Week 0 to Week 3 in MS Quality of Life Inventory (MSQLI) - Mental Health Inventory Scale Score
Description: The Mental Health Inventory (MHI) is an 18-item scale developed as a measure of overall emotional functioning. It is a part of the MS Quality of Life Inventory. The total score is measured from 0-100. The scale is set up so that a higher score indicates better mental health. The change was calculated by taking the Week 3 score and subtracting the Week 0 score. A positive result indicates an improvement in mental health and correlates to a better outcome. A negative result indicates decrease in mental health and correlates to a worse outcome.
Time Frame: Week 0, Week 3
Population: Only 28 subjects completed the study through Wk 7; 2 subjects who discontinued early (AE & withdraw by subject) were active at Wk 3 and were included in the Wk 3 analysis; 14 subjects completed all MHI questions at both the Wk 0 and Wk 3 and were analyzed for this outcome measure. The MHI was added late to the study beginning with subject 22 of 42
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 3 | 6 | 5
units on a scale | -14.8148 (22.8882) | 4.6296 (19.5305) | 4.6667 (6.3050)

52. Secondary Outcome: Change From Week 0 to Week 7 in MS Quality of Life Inventory (MSQLI) - Mental Health Inventory Scale Score
Description: The Mental Health Inventory (MHI) is an 18-item scale developed as a measure of overall emotional functioning. It is a part of the MS Quality of Life Inventory. The total score is measured from 0-100. The scale is set up so that a higher score indicates better mental health. The change was calculated by taking the Week 7 score and subtracting the Week 0 score. A positive result indicates an improvement in mental health and correlates to a better outcome. A negative result indicates decrease in mental health and correlates to a worse outcome.
Time Frame: Week 0, Week 7
Population: Only 28 subjects completed the study through the Wk 7 visit; Of these 28 subjects, only 14 subjects completed all Mental Health Inventory questions at both the Week 0 and Week 7 study visits and were able to be analyzed for this outcome measure. The Mental Health Inventory was added late to the study beginning with subject 22 of 42
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 3 | 5 | 6
units on a scale | -8.8889 (20.3973) | -1.1111 (4.4444) | -8.7037 (23.9487)

53. Secondary Outcome: Change From Week 0 to Week 3 in MS Quality of Life Inventory (MSQLI) - Modified Social Support Scale Score
Description: The Modified Social Support Scale is an 18-item scale developed as a measure of perceived social support. It is a part of the MS Quality of Life Inventory. The total score is measured from 0-100. The scale is set up so that a higher score indicates greater perceived support. The change was calculated by taking the Week 3 score and subtracting the Week 0 score. A positive result indicates an improvement in perceived support and correlates to a better outcome. A negative result indicates a decrease in perceived support and correlates to a worse outcome.
Time Frame: Week 0, Week 3
Population: Only 28 subjects completed the study through the Wk 7 visit; 2 subjects who discontinued early (AE & withdraw by subject) were active at the Wk 3 visit and were included in the Wk 3 analysis; 26 total subjects completed all Modified Social Support scale questions at both the Wk 0 and Wk 3 study visits and were analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 7 | 9 | 10
units on a scale | -6.3988 (19.0288) | 0.2604 (19.1539) | 7.1875 (16.6011)

54. Secondary Outcome: Change From Week 0 to Week 7 in MS Quality of Life Inventory (MSQLI) - Modified Social Support Scale Score
Description: The Modified Social Support Scale is an 18-item scale developed as a measure of perceived social support. It is a part of the MS Quality of Life Inventory. The total score is measured from 0-100. The scale is set up so that a higher score indicates greater perceived support. The change was calculated by taking the Week 7 score and subtracting the Week 0 score. A positive result indicates an improvement in perceived support and correlates to a better outcome. A negative result indicates a decrease in perceived support and correlates to a worse outcome.
Time Frame: Week 0, Week 7
Population: Only 28 subjects completed the study through the Wk 7 visit; Of these 28 subjects, only 26 subjects completed all Modified Social Support scale questions at both the Week 0 and Week 7 study visits and were able to be analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
Number analyzed (Participants) | 7 | 8 | 11
units on a scale | 2.2693 (10.8750) | -4.8177 (21.0544) | -1.4915 (23.0668)

ADVERSE EVENTS:
Time Frame: Adverse event information was collected beginning with the initial dosing visit and continuing through the final follow up visit. Collection period was over approximately 4 months.
Arm/Group | 1) Inhaled Cannabis | 2) Oral THC | 3) Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 3/13 | 1/14 | 0/14
Other Adverse Events (participants affected / at risk) | 13/13 | 14/14 | 12/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1) Inhaled Cannabis (N=13) | 2) Oral THC (N=14) | 3) Placebo (N=14)
hypotension (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
dehydration due to gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
planned insertion of baclofen pump (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
hypersexual thoughts (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1) Inhaled Cannabis (N=13) | 2) Oral THC (N=14) | 3) Placebo (N=14)
euphoria (Psychiatric disorders) | 10 (10) | 6 (6) | 2 (2)
sense of relaxation (Psychiatric disorders) | 3 (3) | 2 (2) | 2 (2)
nausea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 1 (1)
lightheadedness (Cardiac disorders) | 6 (6) | 3 (3) | 0 (0)
dizziness (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1)
difficulty concentrating (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
depression (Psychiatric disorders) | 3 (3) | 4 (4) | 0 (0)
inappropriate laughter (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
headache (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
paresthesia (Nervous system disorders) | 3 (3) | 3 (3) | 3 (3)
paranoia (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0)
sore throat (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
dry mouth (Gastrointestinal disorders) | 2 (2) | 4 (4) | 0 (0)
imbalance (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
generalized weakness (Nervous system disorders) | 2 (2) | 3 (3) | 1 (1)
limb pain (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
upper respiratory infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Multiple Sclerosis relapse (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
hypotension (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
blurred vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
diaphoresis (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
chest pain (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
depersonalization (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
THC dependence (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
flu-like symptoms (General disorders) | 1 (1) | 1 (1) | 0 (0)
dry eyes (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
palpitations (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
visual hallucinations (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
insomnia (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
heightened senses (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
delusions of grandeur (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
hypersexual thoughts (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
drowsiness (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0)
lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
abnormal thinking (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
slurred speech (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
memory problems (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
hematoma on head (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
injury to left arm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
confusion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
facial flushing (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
feeling of heaviness (General disorders) | 0 (0) | 2 (2) | 1 (1)
sensation of cold (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
anorexia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
pre-syncopal episodes (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
"drunk" feeling (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
irritability (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
gastritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
increased difficulty walking (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
increased appetite (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
heartburn (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
tunnel vision (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
headrush (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
hip pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0)
decrease in blood pressure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
itchy throat (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
loquacious (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
influenza (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
polycythemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
pleural effusions (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
renal mass (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
increased fatigue (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
involuntary movement (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
sense of pressure in back of head (General disorders) | 0 (0) | 0 (0) | 1 (1)
back strain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
leg cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
eye irritation (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
dry throat (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
increased stiffness in legs (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
benign tumor left wrist (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated early due to difficulty with enrollment and logistical issues, despite the enrollment period being extended over several years. Data not analyzed due to insufficient enrollment and funds, as well as the departure of the PI.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes